CLINICAL TRIAL: NCT03001180
Title: Identification of Biomarkers for Patients with Vascular Anomalies
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Lymphangiomatosis and Gorham's Disease Alliance (LGDA) (Unknown); Klippel Trenaunay (KT) Support Group (Unknown); CLOVES Syndrome Community Support Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCHMC-LMI
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Vascular Anomaly; Generalized Lymphatic Anomaly; Kaposiform Hemangioendothelioma; Kaposiform Lymphangiomatosis; Gorham-Stout Disease; Klippel Trenaunay Syndrome; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi
Keywords: Generalized Lymphatic Anomaly; Vascular Anomaly; Kaposiform Hemangioendothelioma; Kaposiform Lymphangiomatosis; Vascular Endothelial Growth Factor; Biomarkers; GLA; KLA; KHE; GSD
MeSH Terms: conditions — Vascular Malformations; Kaposiform Hemangioendothelioma; Osteolysis, Essential; Klippel-Trenaunay-Weber Syndrome; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue, Blood, Plasma, and Serum Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will use blood (serum and plasma) and tissue obtained from participants undergoing prescribed surgical resection of vascular anomalies of interest proposed in this study. The study will also use blood (serum and plasma) and tissue collected and stored in a tissue bank maintained by the Department of Hematology/Oncology.

DETAILED DESCRIPTION:
While vascular anomalies are rare diseases, they can be life-threatening and devastating to affected children and their families. Advances in diagnosis, monitoring and therapies will be significantly improved if non-invasive biomarkers that are sensitive and specific can be identified. Obtaining a tissue biopsy to help in diagnosis can actually worsen the disease and so identification of specific blood biomarkers is highly desirable. Studies will measure angiogenic factors in serum and plasma samples at baseline and on therapy. Tissue removed during surgical resection or blood removed prior to sclerotherapy will be used to obtain cells and tissue for the assessment of where biomarkers are coming from and to identify disease-causing pathways for new therapeutic targeting.

ELIGIBILITY:
Inclusion Criteria:

* Any patient having labs drawn as standard of care will have blood drawn for the study if consented/ assented.
* All patients who are undergoing a surgical procedure or sclerotherapy are currently consented for participation in the tissue bank.

Exclusion Criteria:

* N/A

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any participant having labs drawn as standard of care will have blood drawn for the study if consented/assented. All participants who are undergoing a surgical procedure or sclerotherapy are currently consented for participation in the tissue bank. The principle investigator will be looking at tissue from these participants. There is no further recruitment for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-04; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of Biomarkers with Differential Diagnosis | An Average of Every 2 Years
Correlation of Biomarkers with Disease Severity | An Average of Every 2 Years
Correlation of Biomarkers with Response to Therapies | An Average of Every 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy LeCras, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No